CLINICAL TRIAL: NCT03957187
Title: Prevalence and Clinical Associates of Iron Deficiency in Patients With Atrial Fibrillation (AID-AF)
Brief Title: Prevalence and Clinical Associates of Iron Deficiency in Patients With Atrial Fibrillation
Acronym: AID-AF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Koç University (Other)
Collaborators: Vifor Pharma (Industry); Abdi Ibrahim Ilac San. ve Tic A.S. (Industry)
Responsible Party: Sponsor
Other Study IDs: AID-AF 2019
Record Dates: First submitted 2019-03-28; First posted 2019-05-21 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2021-04

CONDITIONS: Iron-deficiency; Atrial Fibrillation
Keywords: iron deficiency; atrial fibrillation
MeSH Terms: conditions — Anemia, Iron-Deficiency; Atrial Fibrillation; Iron Deficiencies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ferritin, iron and iron binding capacity, high sensitive C-reactive protein (CRP) measurement — Ferritin, iron and iron binding capacity will be measured for evaluation of ID using Cobas c-e and Elecsys.
  The relation of inflammation to iron deficiency will be evaluated by high sensitive C-reactive protein measurement.

SUMMARY:
To estimate the prevalence of iron deficiency (ID) in patients with atrial fibrillation

DETAILED DESCRIPTION:
Atrial fibrillation is the most frequent chronic arrhythmia with an increasing prevalence in developed and developing countries. Estimated number of individuals living with chronic atrial fibrillation is 33 million globally. In developed and developing countries, the number of elderly individuals increases steadily and the incidence varies from 0.21 to 0.41/1000 person-years depending on regional differences. Approximately half of atrial fibrillation cases are permanent (chronic), 25% are paroxysmal (ending within one week), and 25% are persistant atrial fibrillation (ending for a week, spontaneous or intervention).

Symptoms and signs of atrial fibrillation vary between individuals, and the clinical picture appears in a wide range of conditions ranging from asymptomatic events to thromboembolic events or patients with severe heart failure. The most common symptoms are; palpitations, fatigue, exercise intolerance, and systemic thromboembolic events in patients who do not receive appropriate anticoagulant treatment. Long-term follow-up, especially in persistent and permanent atrial fibrillation patients results in preserved ejection fraction heart failure and right heart failure. Prevention of thromboembolic events is the most important approach. Patients with paroxysmal, persistent and permanent atrial fibrillation have to take life-long oral anticoagulation therapy if they are at high risk for developing thromboembolic events. In patients with oral anticoagulant therapy, the risk of bleeding increases and hemorrhagic events are seen, ranging from life threatening asymptomatic blood loss to lethal cerebral hemorrhage.

Atrial fibrillation is considered as a chronic inflammatory disease. Both in general population and in patients with cardiac diseases, inflammatory mediators can alter atrial electrophysiology and structure, and thereby increase the tendency to develop atrial fibrillation. Enormous number of studies showed a clear association between inflammatory markers and thromboembolic events in atrial fibrillation.

Anemia is a frequently encountered problem in atrial fibrillation patients with a prevalence of 12.3%. Existing studies suggested an association between anemia and thromboembolic events in atrial fibrillation. However, current evidence supports that it is a marker for increased risk of bleeding after anticoagulant therapy, and two bleeding risk scores (ATRIA and HEAMORRHAGES) included presence of anemia as a component of risk assessment.

Despite of a clear association between anemia and unfavorable events in atrial fibrillation, none of the studies determined the type anemia in these patients so far. In a preliminary single center study, with relatively limited number of cases (n = 101), it is shown that 47.6% of patients with atrial fibrillation had ID according to the criteria used for heart failure patients. B12 (9.9%) and folic acid (12.9%) deficiencies were less frequent Again in the same study, the prevalence of ID was found to be twice as frequent as the paroxysmal atrial fibrillation group in the permanent atrial fibrillation group, suggesting that ID is associated with high sensitive C-reactive protein and N-terminal proBNP levels. The validation of this study findings in a larger, non-retrospective case-group and the clinical determinants of ID in patients with atrial fibrillation will be useful in the clinical evaluation of patients and in planning possible treatment alternatives.

ELIGIBILITY:
Inclusion Criteria:

* Patients with paroxysmal, persistent and permanent non-valvular atrial fibrillation
* Men and women aged over 18 years
* Left ventricular ejection fraction >0.50

Exclusion Criteria:

* Left ventricular ejection fraction <0.50
* Patients with overt symptoms and signs of heart failure
* Patients with a known chronic inflammatory disease
* Patients with hemodynamically significant valvular heart disease
* Patients who had received management for iron deficiency in the preceding 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with atrial fibrillation
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Prevalence of iron deficiency in patients with atrial fibrillation | At enrollment
  To estimate the prevalence of iron deficiency in patients with atrial fibrillation

SECONDARY OUTCOMES:
Assessment of the prevalence of iron deficiency in patients with paroxysmal, persistent and permanent atrial fibrillation | At enrollment
  To estimate the prevalence of iron deficiency in patients with paroxysmal, persistent and permanent atrial fibrillation at enrollment.
Assessment of the relation of iron deficiency to functional capacity | At enrollment
  The functional capacity of the patients will be assessed with 6-minute walk test
Assessment of the relation of iron deficiency to thromboembolic risk score | At enrollment
  Thromboembolic risks will be assessed using CHADSVASC score
Assessment of the relation of iron deficiency to bleeding risk score | At enrollment
  Bleeding risks will be assessed using HASBLED score
Assessment of the relation of iron deficiency to hs-CRP level | At enrollment
  hs-CRP level (milligram/Liter) will be measured in patients with paroxysmal, persistent and permanent atrial fibrillation at enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Ural, Prof., Principal Investigator — Koç University
Locations (1):
- Koc University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided